# **Informed Consent Form**

Protocol Title: Investigator-Initiated, Pilot Study Evaluating the Efficacy of Etanercept in Acute Gout

ClinicalTrials.gov #: NCT03636373

Date: 22 Oct 2020



#### SUBJECT CONSENT TO TAKE PART IN A RESEARCH STUDY

TITLE OF STUDY: Pilot Study Evaluating The Efficacy Of Etanercept In Acute Gout

PRINCIPAL INVESTIGATOR: Naomi Schlesinger, MD

CO-INVESTIGATORS: Robert Eisenstein, MD; Vivien Hsu, MD; Amanda Borham, MD; Ahmed

Abdel-Megid, MD; Dirk F. Moore, Ph.D

This informed consent form provides information about a research study and what will be asked of you if you choose to take part in it. If you have any questions now or during the study, if you choose to take part in it, you should feel free to ask them and should expect to be given answers you completely understand. It is your choice whether to take part in the research. Your alternative to taking part is not to take part in the research.

After all of your questions have been answered and you wish to take part in the research study, you will be asked to sign this informed consent form. You are not giving up any of your legal rights by agreeing to take part in this research or by signing this consent form.

# Who is conducting this research study?

Dr. Naomi Schlesinger, MD is the Principal Investigator of this research study. A Principal Investigator has the overall responsibility for the conduct of the study. However, there are often other individuals who are part of the research team.

Dr. Schlesinger may be reached at The Division of Rheumatology, Department of Medicine, Rutgers - Robert Wood Johnson Medical School, at 125 Paterson Street, New Brunswick, NJ 08901, Phone 732-235-8378.

Dr.Borham may be reached at The Rheumatology Center of New Jersey, 56 Union Avenue Somerville, NJ 08876, Phone 908-280-4495.

The study doctor, Dr. Naomi Schlesinger, MD, or another member of the study team will also be asked to sign this informed consent. You will be given a copy of the signed consent form to keep.

Rutgers, The State University of New Jersey is the Sponsor of this research study. Funding for the study has been provided by Amgen, Inc. The funding will be used to reimburse the Institution for the cost of the study procedures.

#### Why is this study being done?

The study is being done to learn about the effects of the study drug called etanercept for treating the symptoms and pain of an acute attack of gout.

The American College of Physicians recommends that clinicians choose corticosteroids, nonsteroidal anti-inflammatory drugs (NSAIDs), or colchicine to treat patients with acute gout. High-quality evidence showed that corticosteroids, NSAIDs and colchicine are equally effective treatments to reduce pain in patients with acute gout. Corticosteroids should be considered as

10/21/2021

Expiration Date:

first-line therapy in patients without contraindications because they are generally safer and a low-cost treatment option. In this study we will be using the corticosteroid, triamcinolone acetonide 40 mg as our standard treatment and comparing it to etanercept, a new treatment. Triamcinolone acetonide, at a single dose of 40 mg injected intramuscularly (IM), is a popular treatment choice, as it is safe, effective, and offers the potential for treatment with a single dose. We will use triamcinolone acetonide 40 mg IM to compare to a drug called etanercept in this study.

# Why have you been asked to take part in this study?

You are being asked to take part in this study because you have been diagnosed with gout, and you are experiencing an acute gout attack.

# Who may take part in this study? And who may not?

- Males and Females
- Between ages 18 years and 85 years
- With a confirmed history of gout and acute gout attack that started within the past 4 days
- Should be in pain at the time of enrollment in the study

If you are on treatment to lower blood uric acid for at least the past two weeks, you should continue to take the same dose during the study.

The study doctor will review your medications and medical history and decide if you can take part in this study. Also, the study doctor will ask questions about your health. You will not be able to take part in this study if you have a history of alcohol addiction or illegal substance use or abuse. You may not be able to take part in this study if you have a history of rheumatoid arthritis, history of hepatitis B or C, history of active tuberculosis, HIV. Also, if you have an underlying medical condition that is not well controlled at the time of consent. Other conditions that may prevent you from taking part in this study include loss of blood or any serious infections requiring hospitalization in the past 8 weeks, currently pregnant or nursing.

#### How long will the study take and how many subjects will participate?

This study will enroll a total of 40 gout patients from study sites. About 20 subjects will be enrolled at Robert Wood Johnson Medical School and Robert Wood Johnson University Hospital, and another 20 subjects will be enrolled at the Rheumatology center of New Jersey. Your participation will require 4 visits to the study doctor's clinic over about 2 weeks, followed about 2 weeks later by a telephone call. The total study time will be no more than 33 days.

# What will you be asked to do if you take part in this research study?

Study patients recruited at both sites will be asked to do the following study procedures.

| | Visit 1 (Screening and Baseline Study Day 1) | Visit 2<br>(Study Day<br>3-5) | Visit 3<br>(Study Day<br>6-8) | Visit 4<br>(Study Day<br>12-16) | Follow-up<br>phone call<br>(Study Day<br>27-33) |
|---|---|---|---|---|---|
| Informed consent | X | | | | |
| Medical history | Х | | | | |
| Physical exam | Х | Х | Х | Х | |
| Blood work | Х | | Х | | |
| Evaluation | Х | Х | X | Χ | |
| Questionnaires | Х | X | X | X | TITCEDO |

PI: Naomi Schlesinger, MD

| Study medication | x | <b>X</b> (if pain is still severe) | | | |
|---|---|---|---|---|---|
| Screening for side effects | x | x | x | X | x |

#### Study Day 1/Visit 1

If you agree to participate in this study and sign the informed consent, a screening will be performed to see if you can be in the study. This visit includes your medical history, a physical examination, including your height, weight, blood pressure, pulse, and temperature. We will ask you about your demographics (collection of data about yourself like age, gender, and ethnic origin) and about your health including allergies, illnesses and conditions, treatments and operations, general health, and medications you may have taken or may be taking now. Also study nurse will collect your contact information. This will include your name, address and telephone number.

About 2 tablespoons of blood will be collected for testing. These tests include a complete blood count (a test that measures the cells that make up your blood), blood chemistry (a test that measures certain chemicals in blood like sugar and potassium, and helps the doctor to understand how well your organs are working), uric acid (the chemical that helps cause your gout attack), and certain proteins in blood. Also, a urine sample will be collected to determine how well your kidneys are working, and a pregnancy test will be completed if you are a female of child-bearing potential. The study doctor will evaluate your affected joints and determine your overall well-being, and you will complete questionnaires to describe your level of pain and overall well-being.

If you qualify for the study based on your screening, you will be given the study drug. The study is randomized (you will be assigned to one of two treatment groups by chance, like flipping a coin for heads or tails), to decide which treatment you will be given for your gout pain and symptoms.

| Number of patients | Treatment |
|--------------------|--------------------------------------------|
| 20 | Etanercept SC plus Placebo IM |
| 20 | Placebo SC plus Triamcinolone acetonide IM |

Twenty patients will get a single dose of etanercept (the study drug, which is FDA-approved for rheumatoid arthritis, but is not currently approved for gout) 50 mg given subcutaneously (SC; injection under the skin, but not deep enough to enter a vein or muscle) and 20 patients will get a single dose of triamcinolone acetonide (a currently approved treatment for gout) 40 mg given intramuscularly (IM; injection given deep into the muscle). To prevent you or the investigators from knowing which treatment you are given, each patient will also receive a placebo injection (salt water, or normal saline, with no active medication). For example, if you are getting etanercept SC, you will also get the placebo IM, or vice versa.

Rescue medication is a medicine intended to relieve your pain in case you do not sufficiently respond to the study drug. You will be given Tylenol (acetaminophen 500 mg) tablets. You are allowed to take 1 or 2 tablets of Tylenol at a time, every 4 hours if needed. You should not take more than 1 gram (2 tablets of Tylenol) per dose and no more than a total of 3 grams (6 tablets of Tylenol) per day.

You will also be given a prescription for prednisone (20 mg) to take home with you in case your pain is not well controlled by the study medication or Tylenol. If you continue to have pain even


ICF Version and Date 2.1, Mar 10, 2020

IRB ID: Pro2018000562 Approval Date: 10/22/2020 Expiration Date: 10/21/2021

after taking Tylenol, you are allowed to take 20 mg of prednisone by mouth once daily for up to 7 days.

You will also be given a paper diary to take home with you. If you need to take Tylenol (acetaminophen) or Prednisone, you must record the time and the amount taken. At the next study visit, your diary will be reviewed by study personnel.

This visit will take about 6 hours to complete. During this time, you will be completing questionnaires, the study doctor will perform a physical examination and assessments, blood will be drawn, medical and gout history will be collected and study medication will be administered.

# Study Day 4/Visit 2

You will return to the study center 4 days later for Study Day 4/Visit 2. If you are still in pain, you will get a second dose of study drug after evaluation of your pain. You will receive another dose of the same treatment that you received during your first visit.

During this visit, a second physical examination will be conducted. Study investigators will ask you about any side effects of your medication. The study doctor will assess the degree of tenderness and swelling in your affected joint and your overall well-being. The questionnaires describing your level of pain and overall well-being, will be repeated. You will be given the same diary and pain medications to take home as above.

This visit will require approximately 2 hours to complete.

# Study Day 7/Visit 3

You will return to the study center again 3 days later for Study Day 7/Visit 3. This is a follow-up visit only (no more study drug will be given). The same study procedures completed on Visit 2 will be repeated. In addition, about 2 tablespoons of blood will be collected to perform the same tests as Visit 1. You will again be given the same diary and pain medications to take home as above.

This visit will take about 2 hours to complete

# Study Day 12-16/Visit 4

You will return to the study center on Study Day 12-16/Visit 4 for your last follow-up visit, which will include all of the procedures from Visit 2. This will end your use of rescue medications. This visit will take about 2 hours to complete.

# Study Day 27-33

You will receive a follow-up telephone call on Study Day 27-33, to ask about any side-effects you experienced from your medication. This will complete your study participation.

# What are the risks and/or discomforts you might experience if you take part in this study?

#### 1. What are the likely risks with etanercept?

Etanercept may cause all, some, or none of the side effects listed below. These side effects can be mild but could also be serious, life-threatening or even result in death. You may also experience an allergic reaction that has not been seen before.

As of 02 February 2017, approximately 14,595 people have received etanercept in Amgensponsored research studies. Since it was first approved for sale through 02 February 2017, worldwide exposure to etanercept is estimated to be 6,628,257 patient years. Side effects

that other people have had in research studies and with post-marketing use, that are thought to have been caused by etanercept are:

- Very Common side effects (which may affect more than 1 person in 10):
  - a. Injection site reactions—reactions at or near the area of the injection have been seen in other people taking etanercept. Symptoms include redness, tenderness, pain, bruising, warmth, swelling, itching and/or infection at the injection site. These have been reported in subjects receiving etanercept in clinical studies. These reactions usually occurred in the first month (following injection) and disappear in spite of continued etanercept treatment.
  - b. Infections—it is possible that etanercept may make infections worse and that an infection could result in serious illness. Both non-serious and serious infections have been reported in both adults and children in clinical studies, and include viral, bacterial (including tuberculosis), and fungal infections. Infections have been noted in all areas of the body. They have been reported in patients receiving etanercept alone or when used with other drugs that lower your ability to fight infection.
    - Serious infections, such as those that were life threatening, requiring hospitalization and intravenous (IV) antibiotics occur uncommonly (which may affect between 1 and 10 people in every 1000).
    - Serious infections resulting in death have been reported rarely (which may affect between 1 and 10 people in every 10,000).
- Common side effects (which may affect between 1 and 10 people in every 100):
  - a. Allergic reactions—allergic reactions to etanercept have been reported. These reactions may be mild, severe or life-threatening. These reactions may include: headache, flushing, shortness of breath, itching and rash on any part of the body. Hives (itchy raised red bumps on the skin) may develop, or more severe and serious allergic reactions such as dizziness, difficulty breathing, a decrease in blood pressure and/or swelling of parts of the body, the mouth, tongue, and/or throat also occur rarely. Swelling can occur over a period of minutes to several hours after administration of etanercept.
  - b. Development of autoantibodies—after you start taking etanercept, it is possible that your body may make antibodies (proteins that may stop etanercept from working or may cause side effects). Some patients in studies treated with etanercept develop autoantibodies (antibodies that could attach to molecules or substances in the body). Most of the time, these antibodies did not cause problems. Rare cases (which may affect between 1 and 10 people in every 10,000) of a lupus-like syndrome (a disease which has autoantibodies) have been reported.
  - c. Other common side effects include fever.
- Uncommon side effects (which may affect between 1 and 10 people in every 1000):
  - a. <u>Non-melanoma skin cancer</u>—Non-melanoma skin cancers are cancers that form in squamous cells (the top layer of skin cells) or basal cells (the round cells just under the squamous cells). Symptoms of non-melanoma skin cancers may include a change in the appearance of your skin, such as a new growth or a sore that will not heal.

Non-melanoma skin cancers have been reported with etanercept use and are more common in patients with psoriasis. These skin cancers rarely spread to other parts of the body. In clinical studies, patients with psoriasis treated with etanercept, were at a higher risk of getting squamous cell and basal cell skin cancers. Non-melanoma skin

cancers have also been reported uncommonly in patients with rheumatoid arthritis, juvenile idiopathic arthritis, ankylosing spondylitis and psoriatic arthritis.

#### Non-cancer side effects

a. Psoriasis—new psoriasis (patchy kind of skin disease) or worsening of psoriasis (if you already have psoriasis, it may get worse) has been reported in patients during treatment with etanercept. Symptoms may include: scaling red patches or raised bumps which may be filled with a fluid.

#### b. Eve disease

- I. Uveitis (a type of eye inflammation) has been reported with etanercept use. Symptoms may include: in one or both eyes, blurred or cloudy vision, eye redness and/or eye pain especially when looking at bright lights.
- II. Scleritis, a type of eye inflammation affecting the white outer coating of the eye (known as the sclera), can occur in association with rheumatoid arthritis, ankylosing spondylitis and psoriatic arthritis and has been reported with etanercept use. Symptoms may include: in one or both eyes, blurred or cloudy vision, redness in the whites of the eye, eye pain, sensitivity to light and irreversible damage to the eye.
- c. Blood problems—low blood counts have been reported with etanercept use. Reports have included low white blood cells (the cells that help to fight infection), low platelets (the cells that help you to stop bleeding), and low red blood cells (cells that help to carry oxygen to your body). Symptoms of a low blood count may include fever that does not go away, bruising, bleeding, or very pale skin.
- d. Heart failure—congestive heart failure (CHF) (a condition resulting from weakening of the heart muscle) and worsening of CHF in patients who already have it, occurred in patients treated with etanercept. In a clinical trial to treat CHF with etanercept, the results suggested a possible chance that etanercept worsened CHF. Symptoms of heart failure may include shortness of breath and ankle swelling.
- e. Systemic and Cutaneous vasculitis—systemic vasculitis (inflammation of blood vessels in the body) and cutaneous vasculitis (inflammation of blood vessels in the skin) have been reported with etanercept use. Symptoms of vasculitis may include fever, loss of appetite, weight loss, feeling tired, general aches and pains. Systemic vasculitis is uncommon (which may affect between 1 and 10 people in every 1,000). Cutaneous vasculitis is rare (which may affect between 1 and 10 people in every 10.000).
- **f. Elevated liver enzymes**—elevated liver enzymes on blood tests have been reported with etanercept use.
- Rare side effects (which may affect between 1 and 10 people in every 10,000):
  - a. Cancer—There have been reports of cancer in adults, adolescents, and children following etanercept use. It is possible that etanercept may increase the risk of getting lymphoma (cancer of the lymph nodes), leukemia (cancer of the blood) or other cancers. It is unknown if etanercept might influence the development and course of cancer (spreading, the effect of treatment of the cancer, or the cancer coming back after treatment). There have been cases of unusual cancers in children and teenage patients who started using TNF-blocking agents at less than 18 years of age.

Overall cancers occurred in about 1% (1 in 100) of patients with rheumatoid arthritis treated with etanercept in clinical studies for up to 5 years. This is similar to the rate of cancer that would be expected for rheumatoid arthritis or psoriasis patients if they were not receiving etanercept.

RUTGERS | eIRB

IRB ID: Pro2018000562 Approval Date: 10/22/2020

10/21/2021

Expiration Date:

PI: Naomi Schlesinger, MD

# Lymphoma

It is known that subjects with rheumatoid arthritis and psoriasis, whether on etanercept or other treatments, are at a higher risk (up to several times higher) compared with the general population of developing lymphoma (a type of cancer of the lymph nodes). It is also known that those with more active (worse) disease have the highest risk. In rheumatoid arthritis clinical studies, patients treated with etanercept were three times more likely to develop lymphoma than people in general (without rheumatoid arthritis). They were no more likely to develop lymphoma, however, than moderate to severe rheumatoid arthritis patients overall. The role of etanercept and other TNF-blocking therapies in the development of lymphoma is not known.

#### Leukemia

Cases of leukemia have been reported in association with TNF-blocker use. Even in the absence of TNF-blocker therapy, patients with rheumatoid arthritis may have approximately twice the risk of developing leukemia than people without rheumatoid arthritis.

b. Melanoma skin cancer—melanoma (an aggressive form of skin cancer) has been reported in patients taking etanercept. Melanoma develops in the cells that produce melanin which is the pigment that gives your skin its color. The first melanoma symptoms often are a change in an existing mole and/or the development of a new, unusual-looking growth on your skin. Examine your skin so that you become familiar with what your skin normally looks like. This way, you may be more likely to notice any skin changes. Check all areas including those that are hard to see or have someone else check all areas you can't see. Have your doctor do a skin check.

#### c. Non-cancer side effects

- Opportunistic infections—opportunistic infections are unusual infections that occur most commonly when your immune system is weakened.
- Serious skin reactions—severe skin reactions that can be life-threatening rarely occur. These reactions can cause rashes, blistering (on skin, inside the mouth, nose or other areas), and shedding of the skin.
- Nervous system problems— Nervous system events, including multiple sclerosis, convulsions and inflammation of the nerve in the eye, Guillain-Barré syndrome (inflammation of the peripheral nerve in your arms and legs) and inflammation of the spinal cord have been reported in patients taking etanercept. You may experience numbness or tingling, dizziness, weakness in your arms and/or legs, or problems with your vision if you are having a neurologic problem.
- Sarcoidosis—sarcoidosis is a disease that causes inflammation in the lungs and other tissues, and has been reported with etanercept use.
- Other rare side effects—other rare side effects include swelling of the lymph nodes, diarrhea, chest pain, interstitial lung disease (lung scarring), and liver problems such as hepatitis (injury of the liver).
- Very Rare side effects (which may affect less than 1 person in 10,000):
  - a. Blood problems—aplastic anemia (the body stops producing all blood cells) have been reported with etanercept use. Some of the patients with aplastic anemia died. Symptoms of a low blood count may include fever that does not go away, bruising, bleeding, or very pale skin.

#### Other Risks

- a. Inflammatory bowel disease (IBD)—inflammatory bowel disease (is the name of a group of disorders in which the intestines [small and large intestines or bowels] become inflamed, causing redness) has been reported in patients taking etanercept. Symptoms of IBD may include pain in the belly, diarrhea (may be bloody), unexplained weight loss, loss of appetite, bleeding from the rectum, and fever.
- b. Merkel cell skin cancer—Merkel cell skin cancer (an aggressive type of non-melanoma skin cancer) has been reported in patients taking etanercept. Merkel cell cancer affects touch sensitive cells deep in the skin, and often spreads if it is not caught early.

# 2. What are the risks of using etanercept in combination with other drugs?

Tell the study doctor or the study staff about any drugs you are taking, have recently taken, or are planning to take, including herbal remedies, supplements, and drugs you take without a prescription. While we do not know the side effects of using etanercept in combination with all drugs, we do know the following drugs may affect how etanercept works or that etanercept may affect how they work.

- a. Live vaccines should not be given while you are taking etanercept.
- b. Persons with rheumatoid arthritis taking a drug called sulfasalazine with etanercept commonly (which may affect between 1 and 10 people in every 100) had lower numbers of white blood cells (white blood cells help to fight infection). Using these two drugs together could increase your risk of an infection.
- c. Hypoglycemia (low blood sugar levels) has been reported rarely (which may affect between 1 and 10 people in every 10,000) in patients who start taking etanercept and are on medicine for diabetes. Your doctor may need to decrease the dose of your diabetic medication when you start etanercept.
- d. Using a drug called anakinra with etanercept can increase your risk of getting an infection and lower numbers of white blood cells (cells that help to fight infection).
- e. Using a drug called abatacept with etanercept can increase your risk of getting an infection.

Please discuss any concerns you may have with the study doctor.

#### 3. What are the risks of taking the other drugs required by this study?

The following drugs are not being studied by Amgen, but you are required to take them as part of this study. These drugs are often used to treat your condition. The study doctor will talk with you about the risks of taking these drugs.

<u>Triamcinolone acetonide and prednisone are corticosteroids, and can cause any of the following side effects:</u>

- a. High blood pressure;
- b. High blood sugar;
- c. Water retention and weight gain;
- d. Suppression of the adrenal gland, which can cause severe fatigue, depression, weight loss, nausea, vomiting, and diarrhea;
- e. Higher risk of getting a bacterial, viral, or fungal infection, or having reactivation of an old infection such as tuberculosis (TB);
- f. Development or worsening of eye problems such as cataracts or glaucoma;
- g. Development of peptic ulcers, and a higher risk of ulcer bleeding;



- Bone and muscle toxicity, including muscle weakness, tendon rupture, osteoporosis (weakening of bone and increased risk of fracture), and aseptic necrosis of bone (death of bone cells);
- Central nervous system (CNS) toxicity, including headache, insomnia, depression, mood swings, behavior changes, seizures, and tingling or numbness in the fingers or toes.

Acetaminophen is a commonly-used pain medication available without prescription; side effects are not common, but can include:

- a. Upset stomach, vomiting, or stomach pain
- b. Weakness or lightheadedness
- c. Bleeding or unexplained bruising
- d. Allergic reaction (trouble breathing, swelling in the hands, face, lips, mouth, and/or throat, hives, itching, chest tightness)
- e. Liver damage, if taken at too high a daily dose (never take more than 4 grams of acetaminophen per day)
- **4.** What are the risks associated with being pregnant and participating in this study? Pregnant or breastfeeding women, and women planning to become pregnant or planning to breastfeed should not participate in this study as there are risks associated with being pregnant and taking part in this study.

# Could etanercept be harmful to an unborn or breastfed baby?

Taking etanercept during pregnancy or while breastfeeding may involve unknown risks to the unborn or breastfed baby.

Etanercept has been reported to cross (the placenta) from a pregnant mother into the unborn baby. The effects of this on the baby are unknown; however, infants may be at an increased risk of infection. Therefore, the administration of live vaccines to infants for 16 weeks after the pregnant mother's last dose of etanercept is generally not recommended.

Etanercept has been reported to be transferred into breast milk. Babies should not be fed breast milk produced during treatment with etanercept and for an additional 4 weeks after the end of the mother's treatment with etanercept.

#### Triamcinolone acetonide and/or prednisone

There is no evidence in humans that the drug harms the unborn fetus. However, in animal studies corticosteroids have been shown to cause birth defects. Triamcinolone acetonide should only be used during pregnancy when the possible benefits are greater than the risk.

#### Acetaminophen

Acetaminophen is considered safe for use during pregnancy, and is widely used during pregnancy. Results from recent studies suggest a possible association between the use of acetaminophen during pregnancy and subsequent development of attention deficit and hyperactivity disorder (ADHD) in the child. This association has not been proven.

#### **Female Participants**

You and your spouse must use an acceptable method of birth control (unless you are infertile meaning not able to get pregnant or make a female pregnant) throughout the study and for 4

 ICF Version and Date 2.1, Mar 10, 2020

weeks after the last dose of Study Drug. Women should not breastfeed a baby while in this study

If you are unable to become pregnant for one of the following reasons, the use of birth control methods is not required during this study:

- Your healthcare provider has confirmed that you are postmenopausal
- You have had your uterus, or both ovaries, or both fallopian tubes removed

If you could become pregnant, you:

- Should let your sexual partner know you are in this study
- Must agree to practice true sexual abstinence (not have sex) or use an acceptable method(s) of effective birth control during treatment and for an additional 4 weeks after the last dose of etanercept.
- Must discuss your pregnancy prevention method with the study doctor to ensure it is acceptable. You should be aware that true sexual abstinence is the only 100% effective method of birth control.

#### **Birth Control Methods**

Acceptable Methods of Effective Birth Control for Female Participants include:

- Hormonal methods of birth control. Select one option from the following list:
  - o Pills
  - o Implants (placed under the skin by a health care provider
  - Shots/injections
  - Patches (placed on the skin)
- Intrauterine device (IUD)
- Intrauterine hormonal-releasing system (IUS)
- Surgery to tie both fallopian tubes (bilateral tubal ligation/occlusion)
- Your male partner has had a vasectomy and testing shows there is no sperm in the semen.
- Sexual abstinence (not having sex)
- Two barrier methods (one by each partner) and the female partner must use spermicide in addition to a barrier method.
  - The female may select a barrier method from the list below.
  - A female condom is not an option because there is a risk of tearing when both partners use a condom.
    - Diaphragm
    - Cervical cap
    - Contraceptive sponge

#### What if you become pregnant or breastfeed during the study?

If you decide to participate in this study, you must agree to not become pregnant or to breastfeed.

If you are breastfeeding and wish to be in this study, you will be required to discontinue nursing during treatment and for an additional 4 weeks after stopping etanercept.

Since the effect of etanercept is not known, and triamcinolone acetonide is known to cause birth defects in some animals, it is possible that these drugs may cause birth defects. For this reason, no one can be in this study who is pregnant or who could get pregnant while taking the study drug. If you are unwilling to use adequate birth control measures, you should not sign up for this study and are asked not to sign this consent form.

If you think you inadvertently become pregnant, or breastfeed during this study and for an additional 4 weeks after stopping study drug, you must tell the study doctor or study staff right away. Treatment with study drug may be stopped. The study doctor will notify Amgen of the pregnancy or that you are breastfeeding. You will be asked to provide information on the pregnancy or breastfeeding outcome for you and the baby.

# What if your partner becomes pregnant during the study?

If your partner becomes pregnant during treatment and for an additional 4 weeks after stopping etanercept, you must tell the study doctor or study staff right away. The study doctor will notify Amgen of the pregnancy and ask to obtain information on the pregnancy outcome for both the mother and baby.

#### Risks of a blood draw

When your blood is drawn, there may be a bruise, or bleeding, or infection, at the place where your blood is drawn. However, infection is rare.

# Possible interactions between the study drug and other medications

You should not take any over-the-counter medicines, herbal products, vitamins or food supplements while taking part in this study, unless you tell the study doctor and get permission from the study doctor to go on taking these medicines.

There could be additive toxicities if you take non-steroidal anti-inflammatory drugs (NSAIDs) with triamcinolone acetonide. This includes over-the-counter NSAIDs such as ibuprofen (Motrin®), indomethacin (Indocin®), or naproxen (Aleve®). You will follow the instructions of the study doctor about the use of any of these products.

You should also tell the study doctor about all medicines that other doctors may have prescribed for you to take.

# Are there any benefits for you if you choose to take part in this research study?

The benefits of taking part in this study may be an improved control of your gout pain and symptoms. However, it is possible that you may not receive any direct benefit from taking part in this study.

#### What are your alternatives if you don't want to take part in this study?

There are oral anti-inflammatory medications for the treatment of acute gout, including oral colchicine, NSAIDs such as indomethacin, Ibuprofen, or naproxen, and oral corticosteroids such as prednisone or prednisolone. You do not have to participate in this study if you prefer oral treatment over injections. Your alternative is to use these oral options for the treatment of your acute attack and continue your normal treatment for gout, and not to take part in this study.

How will you know if new information is learned that may affect whether you are willing to stay in this research study?

PI: Naomi Schlesinger, MD

During the course of the study, you will be updated about any new information that may affect whether you are willing to continue taking part in the study. If new information is learned that may affect you after the study or your follow-up is completed, you will be contacted.

# Will there be any cost to you to take part in this study?

There is no cost to you for any test or procedure done as part of the study. You will continue to be responsible for any tests or procedures done as part of your normal standard of care.

# Will you be paid to take part in this study?

You can receive a total of \$210 for completing this study. The actual amount you receive is based on the portion of the study you complete. You will receive \$70 for the baseline visit (Visit 1), \$30 for Visit 2, \$70 for Visit 3, \$30 for Visit 4, and \$10 for the follow-up telephone call.

# Who might benefit financially from this research?

- Amgen Inc. (the company developing the study drug) is paying for this research study
- The Study Doctor and the study staff will not profit financially from this study.

# How will information about you be kept private or confidential?

All efforts will be made to keep your personal information in your research record confidential, but total confidentiality cannot be guaranteed.

All of your personal health information, laboratory results, and any other study-related information will be collected and entered into your study records. This information will be securely locked and stored in Rutgers, Robert Wood Johnson Medical School Clinical Research Center or at The Rheumatology Center of New Jersey, and will be available only to study personnel.

The randomization code, which identifies you and the study treatment you are receiving, will be stored on a password-protected computer in the Research Pharmacy in the Clinical Research Center. The Research Pharmacy and the Clinical Research Center will be locked and secured whenever study personnel are not present.

A description of this clinical trial will be available on <u>ClinicalTrials.gov</u>, as required by U.S. law. This website will not include information that can identify you. At most, the website will include a summary of the results. You can search this website at any time.

#### What will happen if you are injured during this study?

Subjects in this study will be exposed to certain risks of personal injury in addition to those associated with standard forms of treatment, which are described in this consent form under "What are the risks and/or discomforts you might experience if you take part in this study?" In addition, it is possible that during the course of this study, new adverse effects of etanercept that result in personal injury may be discovered. The University will make appropriate referrals for medical and/or dental treatment for subjects who sustain personal injuries or illnesses as a direct consequence of participation in the research. The subject's health insurance carrier or other third-party payer will be billed for the cost of this treatment; provided that the University shall not submit to federally funded programs, e.g., Medicare, Medicaid or CHAMPUS, for reimbursement first if submission to such programs is prohibited by law. No financial compensation will be provided by the University and no other type of assistance is available from the University.

What will happen if you do not wish to take part in the study or if you later decide not to stay in the study?

Ruttgers | eIRB

 ICF Version and Date 2.1, Mar 10, 2020

APPROVED

IRB ID: Pro2018000562

Approval Date: 10/22/2020

Expiration Date: 10/21/2021

It is your choice whether to take part in the research. You may choose to take part, not to take part or you may change your mind and withdraw from the study at any time.

If you do not want to enter the study or decide to stop participating, your relationship with the study staff will not change, and you may do so without penalty and without loss of benefits to which you are otherwise entitled.

You may not be able to withdraw your consent for the use of data already collected about you, but if you do not wish to take part, you may withdraw consent from the study at any time. You must do this in writing to Naomi Schlesinger, MD, Department of Rheumatology, Rutgers Robert Wood Johnson Medical School, One Robert Wood Johnson Place, New Brunswick, NJ 08901.

At any time, the study doctor can take you out of this study because it would not be in your best interest to stay in it. Your study doctor can stop treatment even if you are willing to stay in the study.

If you decide to withdraw from the study for any reason, you may be asked to return for at least one additional visit for safety reasons.

# Who can you call if you have any questions?

If you have any questions about taking part in this study or if you feel you may have suffered a research related injury, you can call the study doctor:

Naomi Schlesinger, MD Division of Rheumatology Rutgers Robert Wood Johnson Medical School 732-235-8378

If you have any questions about your rights as a research subject, you can call:

IRB Director (732)-235-9806 New Brunswick/Piscataway

And Human Subject Protection Program 732-235-8578 - New Brunswick

#### What are your rights if you decide to take part in this research study?

You have the right to ask questions about any part of the study at any time. You should not sign this form unless you have had a chance to ask questions and have been given answers to all of your questions.

PI: Naomi Schlesinger, MD

# PERMISSION (Authorization) TO USE OR SHARE HEALTH INFORMATION THAT IDENTIFIES YOU FOR A RESEARCH STUDY

The next few paragraphs tell you about how investigators want to use and share identifiable health information from your medical record in this research. Your information will only be used as described here or as allowed or required by law. If you sign this consent form, you agree to let the investigators use your identifiable health information in the research and share it with others as described below. Ask guestions if there is something you do not understand.

# What is the purpose of the research and how will my information be used?

You are being invited to take part in this research study which is described at the beginning of this form. The purpose of collecting and using your health information for this study is to help researchers answer the questions that are being asked in the research.

#### What information about me will be used?

- All information in your medical record
- Medical history or treatment
- Medications
- Consultations
- Laboratory/diagnostic tests or imaging

# Who may use, share or receive my information?

The research team may use or share your information collected or created for this study with the following people and institutions:

- Rutgers University researchers involved in the study;
- Rheumatology Center of New Jersey researchers involved in the study;
- Robert Wood Johnson University Hospital personnel to communicate information necessary for health care operations;
- The Rutgers University Institutional Review Board and Compliance Boards
- The Office for Human Research Protections in the U.S. Dept. of Health and Human Services
- The Food and Drug Administration
- Amgen Inc. (the company that markets the study drug and is paying for the study)

Those persons or organizations that receive your information may not be required by Federal privacy laws to protect it and may share your information with others without your permission, if permitted by the laws governing them.

#### Will I be able to review my research record while the research is ongoing?

No. We are not able to share information in the research records with you until the study is over. To ask for this information, please contact the Principal Investigator, the person in charge of this research study.

Do I have to give my permission?

No. You do not have to permit use of your information. But, if you do not give permission, you cannot take part in this research study. (Saying no does not stop you from getting medical care or other benefits you are eligible for outside of this study.)

# If I say yes now, can I change my mind and take away my permission later?

Yes. You may change your mind and not allow the continued use of your information (and to stop taking part in the study) at any time. If you take away permission, your information will no longer be used or shared in the study, but we will not be able to take back information that has already been used or shared with others. If you say yes now but change your mind later for use of your information in the research, you must write to the researcher and tell him or her of your decision: Naomi Schlesinger, MD, Department of Rheumatology, Rutgers Robert Wood Johnson Medical School, One Robert Wood Johnson Place, New Brunswick, NJ 08901

# How long will my permission last?

Your permission for the use and sharing of your health information will last until December 31, 2027.

# AGREEMENT TO PARTICIPATE

| 1. Subject consent: |
|---|
| I have read this entire form, or it has been read to me, and I believe that I understand what has been discussed. All of my questions about this form and this study have been answered. I agree to take part in this research study. |
| Subject Name: |
| Subject Signature: Date: |
| 2. Signature of Investigator/Individual Obtaining Consent: |
| To the best of my ability, I have explained and discussed all the important details about the study including all of the information contained in this consent form. |
| Investigator/Person Obtaining Consent (printed name): |
| Signature: Date: |

10/21/2021

Expiration Date: